CLINICAL TRIAL: NCT01495728
Title: Immediate and Short Term Effects of Thoracic Manipulation in Patients With Cervical Radiculopathy
Brief Title: Thoracic Manipulation in Patients With Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spine and Sport, Georgia (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jacki2006
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Radiculopathy; Neck Pain; Manipulation
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrust Manipulation -Thoracic Spine (Experimental): Mid and Upper Thoracic Spine
  Interventions: Procedure: Thrust Manipulation - Thoracic Spine
- Sham Manipulation (Placebo Comparator): Mid and Upper Thoracic Spine
  Interventions: Procedure: Sham Manipulation

INTERVENTIONS:
Procedure: Thrust Manipulation - Thoracic Spine — Mid and Upper Thoracic Spine
  Arms: Thrust Manipulation -Thoracic Spine
Procedure: Sham Manipulation — Mid and Upper Thoracic Spine
  Arms: Sham Manipulation

SUMMARY:
Hypothesis: The group of Cervical Radiculopathy patients receiving thoracic thrust manipulation will demonstrate immediate and short term significant clinically important changes in outcomes when compared to the sham manipulation group.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yrs
* 3 out 4 Items positive of Clinical Prediction Rule for Cervical Radiculopathy

Exclusion Criteria:

* history of previous cervical or thoracic spine surgery
* bilateral upper-extremity symptoms, signs or symptoms of upper motor neuron disease,
* medical "red flags" (e.g., tumor, fracture, rheumatoid arthritis, osteoporosis, and prolonged steroid use).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Global Rating of Change | Pre Treat, Immed, 48-72 hours
  Perceived Improvement
Numeric Pain Rating Scale (Neck & Upper Extremity) | Pre Treat, Immed, 48-72 hrs
  Pain

SECONDARY OUTCOMES:
Neck Disability Index | Pre Treat, Initial, 48-72 hours.
  Disability
Cervical Range of Motion | Pre-treat, immediate post, 48-72 hours
Deep Neck Flexor Endurance | Pre Treat, Immed, 48-72 hours
Numbness and Tingling Scale | Pre Treat, Immed, 48-72 hours
  Rating of distal paresthesia/numbness

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Young, PT, DSc, Principal Investigator — Spine and Sport
Locations (1):
- Spine and Sport, Savannah, Georgia, United States